CLINICAL TRIAL: NCT03422744
Title: Diagnosis of Peripheral Pulmonary Lesions: Benefit of Endoscopic Sample Under Fluoroscopic Controle After Non Contributive Endoscopic Samples Guided by Radial EBUS-miniprobe.
Brief Title: EBUS-Miniprobes Sampling for Peripheral Lung Lesions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough recruitement
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Principal investigator, pneumology, Centre Hospitalier Universitaire Saint Pierre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B076201733056
Record Dates: First submitted 2017-10-06; First posted 2018-02-06 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer; Peripheral Pulmonary Lesions
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with peripheral lung lesion (Experimental): Patient presenting a peripheral lung lesion seen at Ct-scan but invisible at simple endoscopy.
  Intervention : trans bronchial biopsy guided by echo-endoscopic miniprobes.
  Intervention: If first intervention doesn't give a diagnosis we get cytological smear, fine needle biopsy and transbronchial biopsy under fluoroscopic control
  Interventions: Procedure: trans bronchial biopsy guided by echo-endoscopic miniprobes; Procedure: if first one negative: samples under fluoroscopic control

INTERVENTIONS:
Procedure: trans bronchial biopsy guided by echo-endoscopic miniprobes — We get a sample trough transbronchial biopsy guided by echo-endoscopic miniprobe.
Procedure: if first one negative: samples under fluoroscopic control — If no diagnosis with first intervention we get a second sample by cytological smear, fine needle biopsy and transbronchial biopsy under fluoroscopic control

SUMMARY:
There is an interest in characterazing asymptomatic peripheral lung lesions beacause they could be an early form of neoplasm.

These lesions are invisible in the endoscopic exam, so the samples must be made with a guiding technique.

The trans bronchial biopsy after tracking by radial echo-endoscopic miniprobes can be used to collect tissue sample.

When no diagnosis is made with this technique, the attitude can be discussed between different option: follow up versus an other sampling technique (transthoracic ponction, surgery,...).

In this study the investigators will study the interest of a sampling guided by fluoroscopy after a negative sampling guided by radial echo-endoscopic miniprobe.

People presenting with a peripheral lung lesion, invisible with a classical endoscopy, will be included after they sign an informed consent. The bronchoscopy will be executed after a local anesthesia and if there are no visible endobronchial lesions, the radial EBUS mini-probe will be used.

If these samples give an anatomopathologic diagnosis consistent with the clinical context, no other exam will be proposed.

If there isn't a diagnosis after this first exam, a second exam will be proposed to the participants including an histologic smear, a trans bronchial biopsy and a fine needle aspiration under fluoroscopic guidance.

DETAILED DESCRIPTION:
Because of the more frequent use of thoracic imaging by ct-scan, there are a growing number of asymptomatic peripheral lung lesions that are revealed.

As they could be a be an early form of pulmonary neoplasm, it is important for the patient that a definitive diagnosis is made.

These lesions are invisible in the endoscopic exam, so the samples must be made with a guiding technique.

The first guided technique was the biopsy under fluoroscopic control. During the last decade, several other technique have been developed.

Among them is the trans bronchial biopsy after tracking by radial echo-endoscopic miniprobes. This technique has the advantage of needing no exposition to ionizing radiation and lower the risk of pneumothorax, comparing with transthoracic ponction.

In a study made by Guvenc and al. in 2015 this technique achieves a diagnostic in 62 % of the cases.

When the result is negative, the attitude can be discussed between different option: follow up versus an other sampling technique (transthoracic ponction, surgery,...).

In this study the investigators will study the interest of a sampling guided by fluoroscopy after a negative sampling guided by radial echo-endoscopic miniprobe.

Patients presenting with a peripheral lung lesion, invisible with a classical bronchoscopy, will be included after they sign an informed consent. The bronchoscopy will be executed after a local anesthesia and if there are no visible endobronchial lesions, the radial EBUS mini-probe will be used.

If the lesion is spotted, the probe will be withdrawn until the most distal visible carena and the withdrawal distance will be mesured. The biospy forceps will then be introduce at the same distance from this carena and at least five biopsy will be taken.

If these samples give an anatomopathologic diagnosis consistent with the clinical context, no other exam will be proposed.

If there isn't a diagnosis after this first exam, a second exam will be proposed to the participant including an histologic smear, a transbronchial biopsy and a fine needle aspiration under fluoroscopic guidance.

If there is still no diagnosis after this second exam, the attitude will be discussed case by case between a follow up and an other invasive diagnosis mean (transthoracic punction under ct scan control, surgery,…).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting a peripheral lung lesion having given their approval

Exclusion Criteria:

* Lung lesion who according to ct Scan has a greater diameter lesser than 10 mm
* Ground glass lesion
* Lesion that are suspected to be a bronchopneumonia
* Contra-indication for endoscopic exam ( uncontrolled hypoxia, hypercapnia, sympotmatic bronchial hyperreactivity, recent myocardial infarction, heart failure)
* contra-indication for a transbronchial biopsy ( coagulapathy iatrogenic or not, recent uptake of anitaggregant medicines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage Definitive anatomopathological diagnosis | 1 week
  Percentage Definitive anatomopathological diagnosis obtained via the pathological exam of microscopic evaluation, immunostaining and/ or molecular analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD PhD, Principal Investigator — CHU St Pierre
Locations (1):
- CHu Saint Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Endobronchial ultrasound in the management of nonsmall cell lung cancer — https://www.ncbi.nlm.nih.gov/pubmed/23728872
- See also: Computed Tomography Characteristics Predictive for Radial EBUS-Miniprobe-Guided Diagnosis of Pulmonary Lesions — http://www.jto.org/article/S1556-0864%2815%2931655-5/fulltext
- See also: Endobronchial Ultrasound for the Diagnosis of Peripheral Pulmonary Lesions. A Controlled Study With Fluoroscopy — http://www.archbronconeumol.org/en/endobronchial-ultrasound-for-diagnosis-peripheral/articulo/S1579212914001049/